CLINICAL TRIAL: NCT03099083
Title: Real-World Outcome of Psoriasis Patients in Korea on Adalimumab
Brief Title: Real-World Outcome of Psoriasis Subjects in Korea on Adalimumab
Acronym: RAPSODI
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-346
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2019-04

CONDITIONS: Psoriasis
Keywords: Psoriasis; Adalimumab; Humira; Korea
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving adalimumab: Participants with Psoriasis receiving adalimumab

SUMMARY:
The objective of this non-interventional, observational study is to assess the effect of adalimumab on health-related quality of life in participants with Psoriasis in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of Psoriasis by investigator.
* Participant (local definition according to adalimumab label) who is in compliance with eligibility for adalimumab based on the local label.
* Participant must be able and willing to provide written informed consent and comply with the requirements of this study protocol.

Exclusion Criteria:

* Participants who are pregnant or breast feeding at enrolment or wish to become pregnant in the next 24 weeks.
* Participation in any Psoriasis-related clinical trial at the time of enrolment, at baseline or at any point during the study period.
* Participants, who in the investigator's view, may not be able to accurately report their questionnaires

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Psoriasis receiving adalimumab in Korea.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Change in EuroQol 5 dimension (EQ-5D) score up to week 24 | From Week 0 (baseline) to 24
  The EQ-5D measures the subject's overall health state in a descriptive system of health-related quality of life (QoL) states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which can take one of three responses. The responses record three levels of severity ('no problems', 'some problems', and 'extreme problems) within a particular EQ-5D dimension. The EQ-5D results can be converted to health utility scores. Completion time for the EQ-5D is approximately 2-3 minutes.

SECONDARY OUTCOMES:
Change in EuroQol 5 dimension (EQ-5D) score up to week 16 | From Week 0 (baseline) to 16
  The EQ-5D measures the subject's overall health state in a descriptive system of health-related quality of life (QoL) states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which can take one of three responses. The responses record three levels of severity ('no problems', 'some problems', and 'extreme problems) within a particular EQ-5D dimension. The EQ-5D results can be converted to health utility scores. Completion time for the EQ-5D is approximately 2-3 minutes.
Change in PASI score | Week 0 (baseline), Week 16, and Week 24
  PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis).
Percentage of participants achieving Psoriasis Area and Severity Index (PASI) 90 | Up to Week 24
  PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI-90 responders are the participants who achieved at least a 90% reduction (improvement) from baseline in PASI score at Week 24.
Change in EQ-5D Visual Analogue Scale (VAS) | Week 0 (baseline), Week 16, Week 24
  The EQ-5D measures the subject's overall health state in a descriptive system of health-related quality of life (QoL) states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which can take one of three responses. The responses record three levels of severity ('no problems', 'some problems', and 'extreme problems) within a particular EQ-5D dimension. In addition, a VAS rates current health state between 0-100. The EQ-5D results can be converted to health utility scores. Completion time for the EQ-5D is approximately 2-3 minutes.
Percentage of participants achieving Psoriasis Area and Severity Index (PASI) 75 | Up to Week 24
  PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI-75 responders are the participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 24.
Change in Nail Psoriasis Severity Index (NAPSI) score in participants with nail psoriasis | Week 0 (baseline), Week 16, Week 24
  NAPSI grades nails for both nail matrix psoriasis and nail bed psoriasis. The most affected fingernail was determined at Baseline and used for the analysis.
  Nail matrix psoriasis consists of any of the following: pitting, leukonychia, red spots in the lunula, or nail plate crumbling. Nail bed psoriasis is the presence or absence of onycholysis, splinter hemorrhages, oil drop (salmon patch) discoloration or nail bed hyperkeratosis. Scoring for each is based on the following scale:
  * 0 = none;
  * 1 = present in 1/4 nail quadrants;
  * 2 = present in 2/4 nail quadrants;
  * 3 = present in 3/4 nail quadrants;
  * 4 = present in 4/4 nail quadrants.
  The sum of these two scores is the total score for the nail, and ranges from 0 (no nail psoriasis) to 8 (psoriasis in 4/4 nail quadrants).
Change in Short Form (36) Health Survey (SF-36) domain scales | Week 0 (baseline), Week 16, Week 24
  The SF-36 is a subject-reported questionnaire of subject health-related QoL. It measures generic health concepts relevant across age, disease, and treatment groups. There are 36 items in total and the recall period is the last 4 weeks. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. Completion time for the SF-36 is approximately 10 minutes.
Change in Dermatology Life Quality Index (DLQI) | Week 0 (baseline), Week 16, Week 24
  The DLQI is developed as a simple, concise, practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains 10 items dealing with subjects' self-assessments of how their Psoriasis has affected their everyday lives during the latest 7-day period. The DLQI score ranges from 0-30, with 0 corresponding to the best quality of life and 30 the worst. The DLQI has well established properties of reliability and validity when used in a dermatology clinical practice setting.
Percentage of participants achieving Psoriasis Area and Severity Index (PASI) 100 | Up to Week 24
  PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI-100 responders are the participants who achieved at least a 100% reduction (improvement) from baseline in PASI score at Week 24.
Change in subject satisfaction questions | Week 0 (baseline), Week 16, and Week 24
  The Treatment Satisfaction Questionnaire for Medication (TSQM) is a widely used generic measure to assess treatment satisfaction with their medication. This is a 100-point scale with higher scores indicating greater satisfaction with medication and provides scores on four scales - side effects, effectiveness, convenience and global satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (12):
- South Korea (12):
  - Hallym University Sacred Heart Hospital /ID# 161697, Anyang-si, Gyeonggi-do, Gyeonggido
  - CHA Bundang Medical center, CHA University /ID# 161696, Seongnam-si, Gyeonggido
  - Ajou University Hospital /ID# 161698, Suwon, Gyeonggido
  - Yonsei University Health System, Severance Hospital /ID# 166300, Seodaemun-gu, Seoul Teugbyeolsi
  - Hanyang University Seoul Hospi /ID# 169553, Seongdong-gu, Seoul Teugbyeolsi
  - Busan National University Hosp /ID# 166299, Busan
  - Inje University Ilsan Paik Hos /ID# 166302, Goyang
  - Korea University Ansan Hosp /ID# 161695, Gyeonggi-do
  - Korea University Ansan Hosp /ID# 161699, Gyeonggi-do
  - Kyunghee University Hospital /ID# 161694, Seoul
  - National Medical Center /ID# 166298, Seoul
  - Inje University Sanggye Paik H /ID# 166301, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim DH, Son SW, Jeong KH, Ahn J, Lee ES, Kim IH, Lee UH, Park HJ, Ko JY, Kim BS, Kim JJ, Rashid J, Kim KJ. Real-World Outcomes of Adalimumab Treatment for Moderate and Severe Psoriasis in Korean Patients (RAPSODI Study). Ann Dermatol. 2023 Apr;35(2):107-115. doi: 10.5021/ad.22.041. PMID 37041704
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P16-346.pdf